CLINICAL TRIAL: NCT01619098
Title: Evaluating Sequential Strategies to Reduce Readmission in a Diverse Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alison Galbraith (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Cambridge Health Alliance (Other); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Sponsor-Investigator, Alison Galbraith, Assistant Professor, Harvard Pilgrim Health Care
Organization: Harvard Pilgrim Health Care (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R01HS020628 (AHRQ)
Record Dates: First submitted 2012-06-11; First posted 2012-06-14 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Hospital Readmission; Post-discharge Care Transitions; Congestive Heart Failure; Chronic Obstructive Pulmonary Disease
Keywords: Hospital readmission; Care transition; Discharge-transfer intervention; Community health worker; Patient Navigatgor
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive | interventions — Patient Navigation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient Navigator (Experimental): Hospital-based Patient Navigator (a bilingual community health worker) engaged in discharge planning and made outreach phone calls to patients for 30 days after discharge and assisted patints with follow-up appointments, obtaining and taking medications, transportation, financial barriers, and linkages to community resources
  Interventions: Other: Patient Navigator; Other: Usual care
- Usual Care (No Intervention): Home care plan at discharge, outreach phone call from RN at patient's primary care clinic

INTERVENTIONS:
Other: Patient Navigator — In addition to usual care, the intervention adds the services of a community health worker, the Patient Navigator (PN), for study patients. The PN participates in bedside meetings, facilitates communication between the patient and the primary care team, conducts weekly outreach phone calls to further address patient needs, and makes reminder calls prior to all medical appointments to facilitate timely outpatient follow-up.
  Arms: Patient Navigator
Other: Usual care — Usual care includes provision of a Home Care Plan (HCP) to patients at discharge, and electronic transmission of HCP to PCP with telephone follow-up by primary care RN
  Arms: Patient Navigator

SUMMARY:
Hospital readmissions are common, costly, and potentially preventable. They are also potentially responsive to health system interventions. However, it is uncertain which components of care transition interventions are efficacious, for which populations, and at what cost. This randomized controlled study is part of a larger project that will evaluate a three-tiered quality improvement (QI) intervention intended to reduce hospital readmissions within 30 days post-discharge from an urban safety net hospital that serves a racially and linguistically diverse population (the randomized controlled study evaluates Tier 3). Few studies have evaluated care transition interventions to reduce readmissions among low-income, diverse patient populations, and the accumulated evidence on the effects of these multi-faceted interventions on readmission rates has been inconclusive. This project will take advantage of a unique sequence of three QI innovations to reduce hospital readmissions implemented beginning in 2007 in an integrated safety net health care system. The "discharge-transfer" tiers are as follows: 1) Tier 1 includes a comprehensive, individualized home care plan (HCP) reviewed by the medical service floor nurse with the patient prior to discharge; 2) Tier 2 adds the electronic transmission of the HCP to the patient's primary care medical home where, on the business day following discharge, a Registered Nurse makes an outreach telephone call to the discharged patient to confirm comprehension of the HCP and to address medical questions or needs; 3) Tier 3 further adds a community health worker, the Patient Navigator, to participate in bedside discussions to develop rapport and learn about patients' home situations, weekly outreach calls to assess patients' needs and to facilitate communication between the patient and the primary care team, and reminder calls to patients prior to all medical appointments to eliminate barriers to outpatient follow-up. The Aim of the study being registered is to evaluate the effects of an ongoing randomized natural experiment on readmissions, health care use, adherence to medication instructions, and preparedness for discharge. This natural experiment features random assignment to one of two QI interventions, Tier 2 or Tier 3, and exclusively targets patients at high risk for readmission, those with one or more of the following risk factors for readmission: discharge diagnosis of congestive heart failure or COPD; length of stay > 3 days; age > 60; or previous hospitalization within the past six months.

The investigators hypothesize that the Patient Navigator intervention (Tier 3) compared to usual care (Tier 2) will increase the rates of 30-day post-discharge PCP visits; reduce 30-day hospital readmission rates; and reduce the total number of days in hospital in the 180 days following the index admission for high risk patients. The investigators further expect that the PN intervention will improve patient adherence to medication instructions in the HCP and reduce the probability of reported problems with post-discharge care.

ELIGIBILITY:
Inclusion Criteria:

* medical patients discharged to home or skilled nursing facility between October 1, 2011 and June 30, 2013
* Cambridge Health Alliance PCP at time of discharge
* at least one of four risk factors for readmission: discharge diagnosis of CHF or COPD; length of stay >3 days; age >60; or previous hospitalization within the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1510 (Actual)
Dates: Start 2011-10; Primary Completion 2013-06 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Hospital readmission | 30 days
  Inpatient readmission for any reason within 30 days of the index discharge;

SECONDARY OUTCOMES:
Primary and specialty care visit | Number of days to first PCP or specialist visit post-discharge; number of PCP or specialist visits within 7, 15, and 30 days post-discharge
  Number of days to first PCP visit post-discharge; number of days to first PCP or specialist visit post-discharge; number of PCP or specialist visits within 7, 15, and 30 days post-discharge
Emergency department visit | 30 days
  Any ED visit within 30 days post-discharge; Number of ED visits within 30 days post-discharge
Adherence to medication instructions in Home Care Plan | Up to 30 days post-discharge
  A binary indicator of patient adherence to prescription medication instruction in the discharge plan
Patient preparedness for discharge; problems with post-discharge care | Up to 30 days post-discharge
  Satisfaction with inpatient preparation for discharge; receipt of specific written care plan instructions and contact information; satisfaction with understanding of condition, medications, and follow-up appointments; confidence in self-management of post-discharge care; problems with post-discharge care
Costs | within 180 days of discharge
  We will compare the cost per patient of the PN intervention vs usual care from the perspective of Cambridge Health Alliance. Costs will be measured for each patient's 180 days post-discharge and will include Patient Navigator labor, interpreter services, primary care RN labor, and estimated patient care revenues/costs paid for each billable service utilized for study patients using the Medicare fee schedule.
hospital readmission | 15 and 180 days
  Readmission within 15 and 180 days of the index discharge; number of days until first readmission; total number of hospital days in the 180 days post-discharge; readmission before first scheduled PCP or specialist follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Ross-Degnan, ScD, Principal Investigator — Harvard Medical School and Harvard Pilgrim Health Care Institute; Alison Galbraith, MD, MPH, Study Director — Harvard Medical School and Harvard Pilgrim Health Care Institute
Locations (2):
- United States (2):
  - Cambridge Hospital, Cambridge, Massachusetts
  - Whidden Hospital, Everett, Massachusetts

REFERENCES:
- [Derived] Balaban RB, Galbraith AA, Burns ME, Vialle-Valentin CE, Larochelle MR, Ross-Degnan D. A Patient Navigator Intervention to Reduce Hospital Readmissions among High-Risk Safety-Net Patients: A Randomized Controlled Trial. J Gen Intern Med. 2015 Jul;30(7):907-15. doi: 10.1007/s11606-015-3185-x. Epub 2015 Jan 24. PMID 25617166